CLINICAL TRIAL: NCT02109289
Title: Pilot Open-label Study of the Effect of Etanercept on Vascular Inflammation in Patients With Active Rheumatoid Arthritis
Brief Title: Etanercept in Rheumatoid Arthritis and Vascular Inflammation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6032
Record Dates: First submitted 2014-04-03; First posted 2014-04-09 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis; Vascular Inflammation
Keywords: Anti-Tumor necrosis factor alpha; 18-FluoroDeoxyGlucose Positron Emission Tomography; High-sensitivity C- Reactive protein
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methotrexate and Etanercept (Experimental): Patients already taking Methotrexate prior to the study will continue taking 15 mg weekly and start Etanercept 50 mg every week for 16 weeks
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Etanercept is a tumor necrosis factor antagonist
  Other Names: Enbrel

SUMMARY:
The primary goal of this preliminary project is to study the effect of etanercept, a medicine approved by Health Canada for the treatment of rheumatoid arthritis, on the inflammation of certain blood vessels. In particular, the inflammation of the aorta and the carotid arteries will be studied.

This study's goal is to determine if etanercept (that blocks TNF (tissue necrosis factor) alpha) could have an effect on blood vessel inflammation. As well, the information from this study will be used to determine the number of patients to recruit in a future study.

This study will evaluate the effect of etanercept on 10 patients with rheumatoid arthritis at one rheumatology clinic in Montreal. The 10 patients will be recruited at the Montreal Rheumatology Institute (Institut de Rhumatologie de Montréal) and the images of the blood vessels taken at a medical imaging center will be analyzed by the Montreal Heart Institute.

To evaluate vascular inflammation subjects will undergo a PET scan (Positron Emission Tomography).

DETAILED DESCRIPTION:
This study is a 16 week, single center, open label trial, to study the effect of etanercept on vascular inflammation of the ascending aorta and carotid arteries in patients with rheumatoid arthritis (RA).

Patients with active RA already receiving methotrexate for at least 3 months will receive etanercept for 16 weeks. Etanercept will be administered sub-cutaneously using the dose approved in the Canadian product monograph for RA (50 mg every week). Patients will continue methotrexate at a stable dose during the study unless a dose reduction or cessation is required as judged necessary by the study investigator. Positron Emission Tomography (PET) Scan will be performed at baseline and after16 weeks of study treatment with etanercept. At the end of the study, all PET Scan images will be analyzed in a blinded manner by the Montreal Heart Institute core laboratory.

Safety will be assessed using adverse events collection and laboratory hematology and chemistry analysis (screening and Week 4) and pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 to 80 years of age, inclusive.
2. Patient's weight at screening is a maximum of 180 kg.
3. Patient has a clinical diagnosis of active RA for at least 3 months defined as:

   * 2-4 joints with active synovitis OR
   * 1 joint with active synovitis and a high sensitivity C-reactive protein higher than the upper limit.
4. Patient with active synovitis despite treatment for at least 3 months with a dose of methotrexate of at least 15 mg per week.
5. Patient is eligible to receive etanercept according to Canadian Product Monograph.
6. Medications used to control angina, hypertension, serum lipids and any medication that can have an effect on inflammation must be on a stable dose for at least 8 weeks before baseline.
7. Patient with an ascending aorta atherosclerotic plaque inflammation target-to-background ratio of 1.6 or more as determined by 18-FDG uptake measured by PET scanning at pre-enrolment.
8. Female patients of childbearing potential must have a negative serum pregnancy test at the Screening visit.

   Unless patient or patient's partner is in a menopausal state for at least a year, surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation or vasectomy), clinically diagnosed infertile, having a same-sex partner or abstinent,female of childbearing potential or male patient (or his female partner of childbearing potential) is willing to use effective contraceptive method for at least 30 days before Day 0 and at least 4 weeks after the last study drug administration. Effective contraceptive methods are:
   * Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream
   * Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring. Oral contraceptives must have been taken at a stable dose for at least 90 days before study start
   * Intrauterine device (IUD).
9. If result not available in the last 6 months: Patient will be evaluated for latent TB infection with a PPD (Purified Protein Derivative (Mantoux test)) or a Quantiferon Gold test and CXR (chest x-ray).

   Patient who demonstrates evidence of latent TB infection defined below will not be allowed to participate in the study:
   * Either PPD more than or equal to 5 mm of induration or positive Quantiferon Gold, irrespective of Bacillus Calmette-Guerin (BCG) vaccination AND/OR
   * Clinically significant CXR findings or suspicious findings for active TB
10. Patients with diabetes should be well controlled and have a fasting glucose below 11.1 mmol/L.
11. Except for RA, patient is judged to be in good general health as determined by the principal investigator based upon the results of medical history, symptom directed physical examination,laboratory profile,and CXR performed at Screening.
12. Patient must be able and willing to self-administer SC (sub-cutaneous) injections or have a qualified person available to administer SC injections.
13. Patients must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

1. Patient has a history of an allergic reaction or significant sensitivity to constituents of study drug (etanercept), including latex (a component of the pre-filled syringe).
2. Patient has chronic or recurrent infection or history of listeriosis, histoplasmosis or any other invasive fungal or mycobacterial infections, treated or untreated Tuberculosis (TB), persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives drug within 30 days prior to the Day 0 visit or oral anti-infectives within 14 days prior to the Day 0 visit.
3. Patient used any non-biological investigational agents within 30 days or 5 half-lives prior to Day 0 visit (whichever is longer).
4. Patient who has used any biological therapy for the treatment of RA less than 3 months (90 days) or 5 half-lives prior to Day 0 visit (whichever is longer) or patient has received Anakinra/Kineret within the last 2 weeks prior to the Day 0 visit or is likely to receive Anakinra/Kineret during the course of the study.
5. Patient has used a non-biological systemic therapy for the treatment of RA less than 30 days before Day 0, other than methotrexate.
6. Patient is taking or requires oral or injectable corticosteroids at a dose equivalent to more than 5 mg of prednisone daily within 30 days of Day 0 and during the study. Inhaled corticosteroids for stable medical conditions are allowed. Patients taking oral or injectable corticosteroids must be on a stable dose for at least 3 months before Day 0.
7. Patient for whom the treating physician is planning to change the dose of methotrexate or oral corticosteroids during the study.
8. Patient has used a systemic immunosuppressor (eg. Azathioprine, 6-mercaptopurine) less than 30 days before Day 0.
9. Patient who has another musculoskeletal disease that could interfere with or prevent with joint examination
10. Patient who had a myocardial infarction or hospitalization for a cardiac condition within the past 12 weeks.
11. Patient has a pacemaker or a defibrillator.
12. Patient who has a history of acute coronary syndrome, percutaneous coronary intervention, coronary artery dilatation bypass graft, coronary revascularization, carotid endarterectomy, stent installation or carotid revascularization within 12 weeks of baseline.
13. Patient for whom a change in medical treatment for angina, serum lipids, hypertension or any other medication that can have a significant effect on inflammation is planned for the duration of the study.
14. Patient with active or chronic Hepatitis B and /or Hepatitis C.
15. Patient has a known sero-positivity for HIV virus or with or at risk of sepsis syndrome or history of any other immunosuppressive disease.
16. Patient currently uses or plans to use anti-retroviral therapy at any time during the study.
17. Patient has a poorly controlled medical condition, such as uncontrolled diabetes, documented history of recurrent infections, unstable ischemic heart disease, class III or IV (New York Heart Association Functional Classification; NYHA) congestive heart failure, an ejection fraction of less than 30%, recent stroke (within the past 3 months), chronic leg ulcer or any other condition which, in the opinion of the investigator, would put the patient at risk if participating in the study.
18. Patient has lupus erythematosus or history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease (e.g. optic neuritis, visual disturbance, gait disorder/ataxia, facial paresis, apraxia)
19. Patient has history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
20. Female patient who is pregnant or male patient with a pregnant female partner or breast-feeding or considering becoming pregnant during the study or for 4 weeks after the last dose of study medication.
21. Male patient with a female pregnant partner or breast-feeding or considering becoming pregnant during the study or for 4 weeks after the last dose of study medication who is not willing to use effective methods of birth control (a condom or sexual abstinence) during treatment, for the duration of the study and for 4 weeks after the end of treatment.
22. Patient has a history of clinically significant drug or alcohol abuse in the last year.
23. Patient has received a live attenuated vaccine 28 days or less before Day 0 or plan to receive a live attenuated vaccine during the study and up to 4 months after the last study drug administration.
24. Patient with any clinically significant laboratory or exam results judged by the investigator that may put the patient at risk if participating in the study.
25. Patient who plans to travel in an area where tuberculosis is endemic during the study and up to 4 months after the last study drug administration.
26. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Target to background ratio (TBR) from the ascending aorta | 16 weeks
  Change from baseline in target (atherosclerotic plaque) to background (blood) ratio (TBR) from the ascending aorta.

SECONDARY OUTCOMES:
TBR from the mean of both carotid arteries | 16 Weeks
  Change from baseline in the TBR from the mean of both carotid arteries
High Sensitivity C-reactive protein (hsCRP) | 16 weeks
  Change from baseline in hsCRP
Count of swollen and tender joints | 16 weeks
  Change from baseline in swollen and tender joint count
Correlation of TBR from the ascending aorta with hsCRP | 16 weeks
  Correlation between change from baseline in TBR from the ascending aorta and change from baseline in hsCRP
Correlation of TBR from the mean of both carotid arteries with hsCRP | 16 weeks
  Correlation between change from baseline in TBR from the mean of both carotid arteries and change from baseline in hsCRP
Correlation of TBR from the ascending aorta with swollen and tender joint count | 16 weeks
  Correlation between change from baseline in TBR from the ascending aorta at and change from baseline in swollen and tender joint count
Correlation of TBR from the carotid arteries with swollen and tender joint count | 16 weeks
  Correlation between change from baseline in TBR from the carotid arteries and change from baseline in swollen and tender joint count

OTHER OUTCOMES:
Duration of recruitment and recruitment rate | Day 0
Screen failure rate | Day 0
Attrition rate | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Boulos Haraoui, MD, Principal Investigator — Institut de Rhumatologie de Montreal
Locations (1):
- Institut de rhumatologie de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No